CLINICAL TRIAL: NCT00310518
Title: A Phase 2 Multi Center Open Label Study of ARQ 501 in Adult Patients With Recurrent, Persistent or Metastatic Leiomyosarcoma
Brief Title: Safety and Efficacy Study of ARQ 501 in Adult Patients With Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ARQ 501-221
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — beta-lapachone

INTERVENTIONS:
Drug: ARQ 501

SUMMARY:
The purpose of this study is to assess the overall response rate (ORR) of persistent, recurrent or metastatic leiomyosarcoma in patients treated with ARQ 501.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed and dated informed consent prior to study-specific screening procedures.
* Histologically or cytologically confirmed leiomyosarcoma that is persistent, recurrent or metastatic.
* Measurable disease as defined by RECIST.
* Karnofsky performance status >= 70%
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last infusion of ARQ 501.
* Hemoglobin (Hgb) >= 10 g/dL.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1,500/mm3).
* Platelet count >= 100 x 10^9/L (>= 100,000/mm3).
* Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN) or less than or equal to 3.0 x ULN with metastatic liver disease.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN less than or equal to 5.0 ULN with metastatic liver disease.
* Creatinine less than or equal to 1.5 x ULN.

Exclusion Criteria:

* Received three or more prior anticancer chemotherapy regimens.
* Have active, uncontrolled systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment.
* Have received anticancer chemotherapy, immunotherapy, radiotherapy, surgery or investigational agents within four weeks of first infusion.
* Have symptomatic or untreated central nervous system (CNS) involvement.
* Are pregnant or breastfeeding.
* Previous exposure to ARQ 501.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - Premiere Oncology, Santa Monica, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania